CLINICAL TRIAL: NCT05371886
Title: Pharmacokinetics-pharmacodynamics of Morphine With or Without Midazolam Administered by Continuous Infusion in Neonatal Intensive Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PHARAONIC
Record Dates: First submitted 2022-01-31; First posted 2022-05-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Sedation Complication; Mechanical Ventilation in Neonates
Keywords: morphine, midazolam; pharmacokinetics; pharmacodynamics; analgesia; neonates
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The main objective is to estimate a dose-effect relationship of morphine +/- midazolam administration as continuous infusion in neonates undergoing mechanical ventilation through PKPD modelling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-effect relationship of morphine +/- midazolam administration (Other)
  Interventions: Other: Dose-effect relationship of morphine +/- midazolam administration

INTERVENTIONS:
Other: Dose-effect relationship of morphine +/- midazolam administration — Dose-effect relationship of morphine +/- midazolam administration as continuous infusion in neonates undergoing mechanical ventilation through PKPD modelling

SUMMARY:
This study aims to describe a dose-effect relationship of morphine alone and morphine and midazolam administered as continuous infusion in neonates hospitalized in Neonatal intensive care unit and undergoing mechanical ventilation, through PKPD modelling.

DETAILED DESCRIPTION:
This study will include all neonates receiving a sedo-analgesia with continuous infusion of morphine alone or morphine and midazolam during mechanical ventilation in 3 French NICUs. Comfort and pain will be assessed by COMFORTneo pain scores and Newborn Infant Parasympathetic Evaluation Index. Morphine, midazolam and their metabolites' concentrations will be determined on samples taken during a planned blood test. Through PKPD modelling, the dose-concentration-effect relationships will be found and interindividual variability of these drugs in neonates and simulate doses needed to achieve comfort in neonates according to their individual characteristics (gestational age, post-natal age, weight etc.).

ELIGIBILITY:
Inclusion Criteria:

* Neonates < 45 weeks of corrected gestational age
* Hospitalized in a Neonatal Intensive Care Unit
* Undergoing mechanical ventilation
* Patients that receive morphine alone or morphine and midazolam as continuous infusion
* Affiliated to a social security system

Exclusion Criteria:

* Current weight < 600g
* Neonates under palliative care
* Therapeutic hypothermia for perinatal anoxia
* Neonates who underwent a surgical procedure during the past 72 hours
* Neonates receiving concomitantly a paralytic or another drug for sedation or analgesia other than morphine or midazolam (except for paracetamol/acetaminophen)
* Parents refusing that their child participate

Ages: 20 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Effective dose for 50% of patients (ED50 ) of morphine in continuous infusion in neonates ventilated in the neonatal intensive care unit | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  To evaluate which dose is effective, cComfort will be assessed with COMFORTneo score (scale from 6 to 30 with decreasing score with increasing comfort). The dose-response relationship will be assessed with the correlation between a comfortable score (between 11 and 13) and the effective dose for 50% of patients (ED50), by PKPD modeling

SECONDARY OUTCOMES:
Clearance (ml/min/kg) of morphine and midazolam | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  Morphine and midazolam serum levels (mg/L) will be used to describe clearance by PKPD
Volume of distribution (L/kg) of morphine and midazolam | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  Morphine and midazolam serum levels (mg/L) will be used to describe volume of distribution by PKPD modeling
Concentration of morphine | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  Morphine serum levels (mg/L) will be used to describe inter-individual variability by PKPD modeling
Concentration of midazolam | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  midazolam serum levels (mg/L) will be used to describe inter-individual variability by PKPD modeling
Doses of morphine and midazolam (µg/kg/h) | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  PKPD models will be used to simulate doses to determine optimal doses required according to gestational age, postnatal age, corrected age, weight and clinical context
To assess pain responses by the Newborn Infant Parasympathetic Evaluation (NIPE) index | From date of inclusion until the date of end of morphine +/- midazolam treatment, up to 20 weeks
  NIPE Index which provides an observer-independent, quantitative assessment of comfort and analgesia based on analysis of heart rate variability. The NIPE Index ranges from 0 to 100 with increasing index with increasing comfort

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHRU Morvan, Brest
  - CH SUD Francilien, Corbeil-Essonnes
  - CHI Créteil, Créteil
  - CHU Lille, Lille
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No